CLINICAL TRIAL: NCT03828175
Title: Basic Hemodynamics in Correlation With Noninvasive Cardiac Output: A Diagnostic Reliability Issue During Percutaneous Nephrolithotomy Bleeding Under Spinal Anesthesia
Brief Title: Basic Hemodynamic Monitoring Reliability During Percutaneous Nephrolithotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: • MFM-IR.18.03.103 on 5/5/201
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Renal Stone
Keywords: Cardiac output, Hemodynamic, Monitoring, Percutaneous.
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cop variables (Other): non invasive cop vsriables correlation to basic monitoring variables during prone position spinal anesthesia intervention pcnl operation at basic ,1hour and 2hours .
  Interventions: Procedure: spinal anesthesia monitoring

INTERVENTIONS:
Procedure: spinal anesthesia monitoring — After attaching all standard monitors (ECG, NIBP, pulse oximeter) and the COP bio-impedance monitor recording basal data (COP, CI, SV, CPI, Do2, DO2I, SVR, SVV.
  During sitting position intrathecal anesthesia was conducted in the sitting position under complete aseptic condition using heavy bupivacaine 15mg (3ml) plus 10 mic dexamedatomedine 25G needle after 2 ml Lidocaine skin infiltration. lithotomy position till anesthesia level documented T4 and fixed and lower urinary tract endoscopy then shifting the patient to prone position and after adjustment of the prone position precautions 2 bellows one under the chest and one under the pelvis with pliable free moving abdomen jell ring under the patient head knees and in front of heels, then the basal data recording and after that data recording every 10 minutes till end of the operative procedure. Blood sampling at basal, postoperative

SUMMARY:
This prospective pre and post-quasi-descriptive single group interventional study will be done at urology and nephrology center -Mansoura University during the year 2019, for a 3-month duration, starting 1-2-2019 till 1-4-2019 after approval of IRB (Institutional Review Board) code no R/18.03.103 on 5/5/2018, Mansoura Faculty of Medicine. correlating Basic hemodynamics with noninvasive cardiac output for diagnostic reliability during percutaneous nephrolithotomy hidden bleeding under spinal anesthesia

DETAILED DESCRIPTION:
Hypothesis: On the concept of patient safety, using basic noninvasive monitoring tools (Blood pressure, HR, pulse oximetry O2 Saturation) are late and deceiving and non-reliable hemodynamic measuring tools in diagnosing the progression of the silent hidden bleeding during percutaneous nephrolithotomy surgery (PCNL) operations and necessitate adding noninvasive COP (bioimpedance based) monitor for minute to minute detection of the hemodynamic changes during (PCNL) surgery (necessitates high level spinal anesthesia and prolonged prone position with its hemodynamic burden, carries high risk of inaccessible uncontrollable bleeding).

The aim of the work:

Targeting more intraoperative patient safety by determination of the credibility of basic hemodynamic monitors in reflecting the real cardiopulmonary functions during PCNL operation (high risk is hidden bleeding) under prone position spinal anesthesia.

Achieved by using correlation between intraoperative noninvasive thoracic bioimpedance [COP -oxygenation] monitor and the usually used basic intraoperative [hemodynamic-oxygenation] monitoring systems; two outcome categories will be correlated; a)-Circulatory category: thoracic bioimpedance based COP hemodynamic parameters including (cardiac output COP-stroke volume SV -stroke index SI- cardiac index CI-cardiac performance index CPI-stroke volume variability SVV, systemic vascular resistance SVR, systemic vascular resistance index SVRI) correlation with the usual basic hemodynamic monitoring dependent parameters noninvasive blood pressure NIBP (systolic SBP and mean MAP) and the heart rate HR. b)- Oxygenation category: (Oxygen delivery (Do2), Oxygen delivery index (Do2I), correlation with the basic monitor pulse oximeter oxygen saturation (Sao2).

Correlation will be done at 3 times first basal (just after prone position adjustment and before PCNL puncture, after 60 min then after 120 minutes of prone position adjustment.

Patient & Methods:

This prospective pre and post-quasi-descriptive single group interventional study will be done at urology and nephrology center -Mansoura University during the year 2019, for a 3-month duration, starting 1-2-2019 till 1-4-2019 after approval of IRB (Institutional Review Board) code no R/18.03.103 on 5/5/2018, Mansoura Faculty of Medicine.

Sample size calculation Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 15.0.5 for Windows (2017) using results obtained by a pilot study conducted on 5 patients at Mansoura urology and nephrology center (January-2019) with the difference in reliability (as measured by Cronbach's alpha) between mean non-invasive blood pressure (MAP) and stroke volume index (SVI) as the primary outcome. We choose the SVI over other monitoring tools as cardiac output or the cardiac index due to its relatively more available measurement tools. A sample size of 32 patients is needed to achieve 90% power and detect the difference between the Cronbach's alpha of the MAP (considered to be the null hypothesis) of 0.974 and the Cronbach's alpha for the SVI of 0.988 using a two-sided F-test with a significance level of 0.05. The expected number of drop-outs is 8, so a total of 40 patients will be enrolled into the study.

Preparation:

After patient examination and consultation about any comorbidities. Consent will be taken after explanation of the anesthetic procedures, 1000 ml Ringers solution during 30 minutes before anesthesia the morning of the procedure.

Intraoperative management:

After attaching all standard monitors (ECG, NIBP, pulse oximeter) and the COP bio-impedance monitor recording basal data (COP, CI, SV, CPI, CaO2, Do2, DO2I, SVR, SVV.

During sitting position intrathecal anesthesia was conducted in the sitting position under complete aseptic condition using heavy bupivacaine 15mg (3ml) plus 10micrograms dexamedatomedine using 25G needle after 2 ml Lidocaine skin infiltration. lithotomy position till anesthesia level documented T4-5 and fixed and lower urinary tract endoscopy then shifting the patient to prone position and after adjustment of the prone position precautions 2 bellows one under the chest and one under the pelvis with pliable free moving abdomen jell ring under the patient head knees and in front of heels, then the basal data recording and after that data recording every 10 minutes till end of the operative procedure,With basal& postoperative HB detection.

Episodes of perioperative: Hypotension is defined as mean arterial blood pressure (MBP) less than 65 mmHg, will be managed by using bolus doses of ephedrine 6 mg, fluids and blood transfusion according to patients HB level with blood transfusion cut point of 8mg/dl. Bradycardia is defined as HR less than 60 b/m. will be managed by atropine 0.5 mg bolus. Desaturation is defined as SaO2< 90% will be managed by stop surgery, increase O2 flow via the oxygen face mask from 5 to 10 liters/minute, chest auscultation and verbal patient examination with shift to lithotomy position if desaturation persist and keep all tools and drugs ready for intubation and mechanical ventilation if needed. Nausea will be managed by treatment of hypotension as a common cause and propofol 20 mg. vomiting will be treated by dexamethasone 0.1mg/Kg with metoclopramide 0.1mg/Kg.

Intraoperative pain will be managed by fentanyl 0.5 mcg/kg, IV infusion of paracetamol 10mg/kg, propofol 50 mg increments, or general anesthesia using ETT and inhalational maintenance if there is still more than 15 min expected time to end the surgical procedure by shifting to lithotomy position and then General anesthesia induction with endotracheal intubation with mechanical ventilation then continue surgery and the case excluded from the study and replaced as a dropout case.

Primary outcome:

Stroke volume index (SVI)

Secondary outcome:

Hemoglobin (HB) (basal prior surgery &Postoperative), cardiac output (COP)- Stroke volume (SV)- Cardiac performance index (CPI)-systemic vascular resistance (SVR) - systemic vascular resistance index (SVRI) - stroke volume variability (SVV)- Oxygen delivery DOI-cardiac Index-Oxygen delivery (DO2)- Oxygen delivery index (DO2I). Noninvasive Intraoperative hemodynamic (systolic blood pressure (SBP), mean blood pressure (MAP), heart rate (HR) and O2 saturation (SaO2). All mentioned variables will be recorded basal and every 10 minutes till end of surgery.

Statistical analysis

IBM's SPSS statistics (Statistical Package for the Social Sciences) for Windows (version 25) will be used for statistical analysis of the collected data. Shapiro-Wilk test will be used to check the normality of the data distribution. Normally distributed continuous variables will be expressed as mean ± SD while categorical variables and the abnormally distributed continuous ones will be expressed as a median and inter-quartile range or number and percentage (as appropriate). Reliability analysis will be conducted using Cronbach's alpha test. Student t-test and Mann-Whitney will be used for normally and abnormally distributed continuous data respectively. Chi-square test will be used for categorical data using the crosstabs function. All tests will be conducted with 95% confidence interval. If needed, bivariate correlations will be assessed using Pearson's or Spearman's correlation coefficient depending on the nature of data. P (probability) value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for percutaneous nephrolithotomy endoscopic operation
2. ASA I-III.
3. Both sexes,
4. Age 18 - 70 years.
5. PCNL operation time ≥120 minutes.

Exclusion Criteria:

1. Patient refusal.
2. PCNL operation time <120 minutes.
3. Hypersensitivity to amide local anesthetics.
4. General contraindications to spinal anesthesia, coagulopathy.
5. Cardiac, hepatic, renal or respiratory failure.
6. Difficult communication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Stroke volume index (SVI) | up to 120 minutes.
  continuous stroke volume index (stroke volume divided by the body weight) during prone position spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Faculty of Medicine, Al Mansurah, DK, Egypt